CLINICAL TRIAL: NCT06918808
Title: A Phase 2a Study of Allogeneic Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicle Isolate Product (DB-3Q) in Patients With Perianal Fistulizing Crohn's Disease
Brief Title: DB-3Q bmMSC-EVs in Patients With Perianal Fistulizing Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3Q-PFCD-201
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Perianal Fistula Due to Crohn's Disease

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled, sequential cohort, ascending dose clinical trial to evaluate the safety and determine the efficacy of ascending doses of DB-3Q for the treatment of PFCD.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Single dose DB-3Q 15 mL direct injection (Experimental)
  Interventions: Biological: DB-3Q
- Single dose Placebo 15 mL direct injection (Placebo Comparator)
  Interventions: Biological: Placebo
- Single dose DB-3Q 30 mL direct injection (Experimental)
  Interventions: Biological: DB-3Q
- Single dose Placebo 30 mL direct injection (Placebo Comparator)
  Interventions: Biological: Placebo
- Single dose DB-3Q 15 ml IV and DB-3Q 30 mL direct injection (Experimental)
  Interventions: Biological: DB-3Q
- Single dose Placebo 15 ml IV and Placebo 30 mL direct injection (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DB-3Q — DB-3Q (IMP) is the frozen liquid formulation of acellular secretome proteins and extracellular vesicles isolated from human bmMSC and processed under current Good Manufacturing Process standards.
  Arms: Single dose DB-3Q 15 mL direct injection; Single dose DB-3Q 15 ml IV and DB-3Q 30 mL direct injection; Single dose DB-3Q 30 mL direct injection
Biological: Placebo — 0.9% NaCl
  Arms: Single dose Placebo 15 mL direct injection; Single dose Placebo 15 ml IV and Placebo 30 mL direct injection; Single dose Placebo 30 mL direct injection

SUMMARY:
This is a double-blind, randomized, placebo-controlled, sequential cohort, ascending dose clinical trial to evaluate the safety and determine the efficacy of ascending doses of DB-3Q for the treatment of Perianal Fistulizing Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from participant
2. Men and women 18-75 years of age with a diagnosis of Crohn's Disease for at least six months duration prior to Day 1
3. Single and/or multi-tract perianal fistula(s) with 2 or fewer openings, that are actively draining
4. Failed at least one medical therapy within the last year including, but not limited to, antibiotics, immunomodulators (6-MP, methotrexate, azathioprine), monoclonal antibodies (adalimumab, certolizumab, golimumab, guselkumab, infliximab, risankizumab, ustekinumab, vedolizumab), or small molecule inhibitors (tofacitinib, upadacitinib)
5. Previous failed surgical intervention, including seton placement at least two weeks prior to screening, or are not candidates for surgical intervention or are not willing to undergo surgical intervention for the management of their fistula
6. Medical therapy for CD stable for at least 2 months prior to Day 1 (Changes in dosing or dosing intervals related to serum drug levels are not permitted)

Exclusion Criteria:

1. Lack of informed consent
2. Pregnant woman, woman of childbearing potential without a documented negative urine or serum pregnancy test, or woman who is breast feeding
3. A participant who is unwilling to use medically acceptable contraception methods during participation in study
4. Active perianal abscess or infection at screening or Day 1
5. Clinically significant medical conditions within six months before Day 1 that would, in the opinion of the Investigator, compromise the safety of the participant
6. Confirmed HIV, Hepatitis B, or Hepatitis C infections
7. History of cancer including melanoma (with the exception of localized non-melanoma skin cancers) within one year of screening
8. History of colorectal cancer within 2 years of screening
9. Use of investigational therapy or treatment within 30 days prior to Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Combined Remission | 24 Weeks
  Clinically confirmed 100% closure of all treated external openings, without development of new fistulas or abscesses and drainage > 1 cm by the external openings, occurring spontaneously or after gentle finger compression; and on blinded central review of the MRI results, combined imaging endpoint of >50% reduction in MAGNIFI-CD score and >20% increase in perianal fistula fibrosis-to-fluid ratio.

SECONDARY OUTCOMES:
Combined Remission | 12 Weeks
  Clinically confirmed 100% closure of all treated external openings, without development of new fistulas or abscesses and drainage > 1 cm by the external openings, occurring spontaneously or after gentle finger compression; and on blinded central review of the MRI results, combined imaging endpoint of >50% reduction in MAGNIFI-CD score and >20% increase in perianal fistula fibrosis-to-fluid ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center/NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IP protection